CLINICAL TRIAL: NCT00435955
Title: MULTICENTER RANDOMIZED PROGRAM COMPARING HIGH-DOSE CHEMOTHERAPY + RITUXIMAB AND PERIPHERAL BLOOD PROGENITOR CELL (PBPC) AUTOGRAFT vs. CHOP + RITUXIMAB AS FIRST-LINE TREATMENT FOR PATIENTS WITH HIGH-RISK FOLLICULAR LYMPHOMA
Brief Title: Comparison of High-Dose Chemotherapy + Rituximab and CHOP + Rituximab in High-Risk Follicular Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Collaborators: University of Turin, Italy (Other); Gruppo Italiano Trapianto di Midollo Osseo (Other); Gruppo Italiano Studio Linfomi (Other); Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3320
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2007-02-16 (Estimated); Status verified 2007-02

CONDITIONS: Follicular Lymphoma
Keywords: Follicular lymphoma; age adjusted IPI >1; IIL score > 2; Molecular remission; High dose chemotherapy and autologous transplantation; Rituximab
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Drug Therapy; Transplantation, Autologous; Rituximab

INTERVENTIONS:
Procedure: High dose chemotherapy with autologous transplantation
Drug: Rituximab

SUMMARY:
The purpose of this study is to determine whether an intensified treatment plus Rituximab followed by autologous transplantation is superior to a conventional chemotherapy regimen also supplemented with Rituximab.

DETAILED DESCRIPTION:
The place of intensified regimens with autologous stem cell transplantation (ASCT) is poorly defined in FL at diagnosis . Most data arise from studies performed in the pre-Rituximab age. According to these studies, ASCT improved overall survival versus standard salvage approaches in relapsed patients with a high proportion of patients achieving a durable molecular remission. Data at diagnosis are less clear. Three studies have been so far published with contradictory results. Two of these studies showed that intensive therapy ensures a better disease control although in one study a significant extra-mortality from secondary tumors was observed in the intensified arm. A third study found no advantage for patients treated intensively. These results led to the widespread notion that ASCT is not superior to conventional chemotherapy in unselected FL patients. Our previous non-randomized experience employing high dose sequential chemotherapy with a final TBI-free ASCT added some clues to these considerations. Our study employs an autografting procedure which is associated to fewer secondary tumors as it does not include total body irradiation. Moreover we have observed that the our regimen (named HDS) is particularly effective in high-risk patients, suggesting that this specific subgroup is the most appropriate setting for intensified regimens

The present multicenter open label randomized trial took advantage of these observations. In addition we have included Rituximab in both arms as the inclusion of this novel agent is expected to significantly modify the performance of available treatments. We have thus compared a Rituximab-supplemented version of HDS (R-HDS) regimen with six CHOP courses supplemented by an identical number of Rituximab courses. Aim of the study was verify if an intensified approach could be beneficial as first line treatment of high-risk FL patients in the Rituximab age.

ELIGIBILITY:
Inclusion Criteria:

1. Follicular Lymphoma at diagnosis
2. Stage >I
3. age-adjusted I.P.I. score 2 or 3 or three or more adverse factors of the I.L.I. score

Exclusion Criteria:

1. Serum positivity for HIV, HCV. HBsAg-positive only if active viral replication, assessed by HBV-DNA was present.
2. Major alterations of heart, lung, kidneys, liver, except for those directly disease-related;
3. Evidence of second tumors;
4. Previous chemotherapy( except patients who received limited radiotherapy);
5. Cerebral or CNS involvement.
6. Drug addiction or severe psychiatric disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240
Dates: Start 2000-03

PRIMARY OUTCOMES:
Event free survival at three years

SECONDARY OUTCOMES:
Overall survival
CR rate
Progression free survival
Disease free survival I
Incidence of secondary myelodisplasia and solid cancer
Rate of molecular remission
Predictive value of molecular remission

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tarella, MD, Principal Investigator — Università di Torino, Azienda Ospedaliera San Giovanni Battista; Marco Ladetto, MD, Principal Investigator — Università di Torino Azienda Ospedaliera San Giovanni Battista; Alessandro Pileri, MD, Principal Investigator — Università di Torino Azienda Ospedaliera San Giovanni Battista (Now retired); Mario Boccadoro, Principal Investigator — Università di Torino/Azienda Ospedaliera San Giovanni Battista B; Alessandro Gianni, Principal Investigator — Istituto Tumori di Milano, Milano Italy
Locations (1):
- Divisione di Ematologia Universitaria, Torino, Italy

REFERENCES:
- [Derived] Ladetto M, De Marco F, Benedetti F, Vitolo U, Patti C, Rambaldi A, Pulsoni A, Musso M, Liberati AM, Olivieri A, Gallamini A, Pogliani E, Rota Scalabrini D, Callea V, Di Raimondo F, Pavone V, Tucci A, Cortelazzo S, Levis A, Boccadoro M, Majolino I, Pileri A, Gianni AM, Passera R, Corradini P, Tarella C; Gruppo Italiano Trapianto di Midollo Osseo (GITMO); Intergruppo Italiano Linfomi (IIL). Prospective, multicenter randomized GITMO/IIL trial comparing intensive (R-HDS) versus conventional (CHOP-R) chemoimmunotherapy in high-risk follicular lymphoma at diagnosis: the superior disease control of R-HDS does not translate into an overall survival advantage. Blood. 2008 Apr 15;111(8):4004-13. doi: 10.1182/blood-2007-10-116749. Epub 2008 Jan 31. PMID 18239086